CLINICAL TRIAL: NCT05392179
Title: An Open-label, Phase II Study of ADX-2191 in Subjects With Retinitis Pigmentosa
Brief Title: A Study in Subjects With Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADX-2191-RP-001
Record Dates: First submitted 2022-03-28; First posted 2022-05-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Retinitis Pigmentosa
Keywords: ADX-2191; Methotrexate; Retinitis Pigmentosa; Rhodopsin Mutation P23H
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-2191 Three Injections (Experimental)
  Interventions: Drug: ADX-2191
- ADX-2191 Six Injections (Experimental)
  Interventions: Drug: ADX-2191

INTERVENTIONS:
Drug: ADX-2191 — Monthly intravitreal injections of ADX-2191 (400 µg in 0.05 mL) for a total of three injections. Evaluation through week 16.
  Arms: ADX-2191 Three Injections
Drug: ADX-2191 — Monthly intravitreal injections of ADX-2191 (400 µg in 0.05 mL) for a total of six injections. Evaluation through week 16.
  Arms: ADX-2191 Six Injections

SUMMARY:
An open-label Phase II clinical trial, 8 (eight) subjects with retinitis pigmentosa due to rhodopsin mutations (including P23H) will be identified and treated with serial intravitreal injections of ADX-2191 in the worse seeing eye. Ocular structure and function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Up to 8 adult patients age 18 or older
2. Diagnosis of retinitis pigmentosa due to rhodopsin gene mutation, including P23H
3. Impairment on Visual Field as determined by perimetry

Exclusion Criteria:

1. Age < 18 years
2. Pregnant
3. Previous inflammatory/infectious events involving the eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | 16 weeks
  Assessing the safety of ADX-2191 in patients with retinitis pigmentosa from AE collection

SECONDARY OUTCOMES:
Change in visual acuity | 16 weeks
  Assessing the change in visual acuity in patients with retinitis pigmentosa treated with ADX-2191 using the Early Treatment Diabetic Retinopathy (ETDRS) chart.
Central retinal sensitivity | 16 weeks
  Assessing the central retinal sensitivity in patients using microperimetry, measured in decibels
Change in dark-adapted retinal sensitivity | 16 weeks
  Assessing the change in dark-adapted retinal sensitivity in patients using dark adapted chromatic perimetry, measured in decibels
Assessment for change in central subfield foveal thickness and ellipsoid zone area/width | 16 weeks
  Assessing the change in central subfield foveal thickness and ellipsoid zone area/width in patients using Spectral-Domain Optical Coherence Tomography (SD-OCT) as measured in square millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No